CLINICAL TRIAL: NCT06273254
Title: A Bioequivalence Study of Two Formulations of Sacubitril/Valsartan 49 mg/51 mg Film-coated Tablets in Healthy Thai Subjects Under Fasting Conditions
Brief Title: A Bioequivalence Study of Sacubitril/Valsartan Film-coated Tablets Under Fasting Conditions
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Viatris Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: SCVL-TFZ-1009
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Bioequivalence Study
MeSH Terms: interventions — sacubitril; Valsartan; sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product (Experimental): Sacubitril and Valsartan Tablets 49mg/51mg to be orally administered
  Interventions: Drug: Sacubitril and Valsartan Tablets 49mg/51mg
- Reference product (Active Comparator): Entresto® (48.6 mg sacubitril and 51.4 mg valsartan as sodium salt complex) to be orally administered
  Interventions: Drug: Entresto® (Sacubitril and Valsartan Tablets 49mg/51mg)

INTERVENTIONS:
Drug: Sacubitril and Valsartan Tablets 49mg/51mg — Each tablet contains Sacubitril 49 mg and Valsartan 51 mg
  Arms: Test Product
Drug: Entresto® (Sacubitril and Valsartan Tablets 49mg/51mg) — Each tablet contains 48.6 mg sacubitril and 51.4 mg valsartan as sodium salt complex
  Arms: Reference product

SUMMARY:
Primary objective is to is to evaluate the bioequivalence of two formulations

DETAILED DESCRIPTION:
To evaluate the bioequivalence of two formulations of sacubitril/valsartan 49 mg/51 mg film coated tablets, Entresto® (Reference) and Sacubitril and Valsartan Tablets 49mg/51mg (Test), after a single oral dose administration in healthy Thai subjects under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

1. Thai Male/Female must be 18-55 years of age, body weight > 50.0 kg with body mass index (BMI) = 18.0-30.0 kg/m2, inclusive.
2. Must be in good health as determined by medical history, vital signs (blood pressure (systolic blood pressure not lower than 100 or not over 139 mmHg, diastolic blood pressure not lower than 70 or not over 89 mmHg), body temperature, pulse rate, respiratory rate) and physical examination or showing no clinically significant abnormalities in the opinion of Principal/Clinical Investigator or designated physicians
3. Screening ECG without clinically significant abnormalities
4. Screening visit laboratory values of blood test including hematology (CBC with differential), FBS (Fasting Blood sugar), BUN (Blood urea Nitrogen), Cr, and liver function test (AST (Aspartate transaminase), ALT (Alanine transaminase) , total bilirubin and ALP (Alkaline phosphatase) must be within the normal range or showing no clinically significant abnormalities in the opinion of Principal/Clinical Investigator or designated physicians.
5. Urinalysis results within normal limit or showing no clinically significant abnormalities in the opinion of Principal/Clinical Investigator or designated physicians.
6. Must have serum HBsAg, anti-HCV and anti-HIV negative
7. Female subject must have serum β-hCG negative or showing no clinically significant abnormalities in the opinion of Principal/Clinical Investigator or designated physicians.
8. Subject willing to avoid or follow precautions while driving, operating machinery and while working on high elevations.
9. Female subject of childbearing potential or male subject agrees to use an acceptable birth control method from screening visit to the followup visit. The acceptable birth control method is defined as a barrier method of contraception (including condoms, intrauterine device and diaphragm with spermicidal agent) or total abstinence from sexual intercourse from visit 1 to the follow-up visit. Hormonal contraceptives are not acceptable.
10. Female subject of non-childbearing potential (hysterectomy, both ovaries removed, surgically sterilized or postmenopausal (for at least 12 consecutive months of amenorrhea))
11. Female subject must agree not to become pregnant for the entire participation period and must have a negative result for a urine pregnancy test performing prior to dosing at Period 1, Period 2, Period 3 and Period 4.
12. Non-smoker (never smoked or no smoking within the previous 1 year)
13. Subject willing to not participate in blood donations (≥500 mL) until 56 days after completion of the study (last subject visit) and willing to not participate in clinical research studies until 30 days after completion of the study (last subject visit).
14. Refrain from using herbal medications, cannabis containing products, dietary supplements (e.g., St. John's Wort, ginkgo biloba, garlic supplements), vitamins, grapefruit or grapefruit juice, or pomelo within 14 days before the first administration of investigational product (Day 1). Subjects must agree to refrain from these items until the last collection time-point of Period 4.
15. Subject must have ended any systemic medications or any medications that have any impact on gastrointestinal system at least 30 days prior to Day 1 or at least 5 times of elimination half-life prior to Day 1 and agree to continue their refraining throughout the follow-up period.
16. Subject must refrain from drinking caffeine and alcohol for at least 48 hours prior to Day 1 and agree to continue their refraining throughout the last collection time-point of Period 4.
17. Have the ability to understand the requirements of the study and must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

1. Known hypersensitivity to sacubitril or valsartan or any other similar class of drugs or its components
2. Past medical history of renal and hepatic insufficiency
3. Subject has a history of any illness that, in the opinion of Principal/Clinical Investigator or designated physicians, might confound the result of the study or pose an additional risk in administering investigational product to the subject. This may include but is not limited to: a history of relevant drug or food allergies; history of cardiovascular, gastrointestinal, central nervous system disease, renal and hepatic impairment; history or presence of clinically significant illness; or history of mental illness that may affect compliance with study requirements.
4. History of hereditary or idiopathic angioedema
5. Have a history of angioedema related to previous ACE inhibitor or ARB therapy
6. Have history of drug abuse (in the opinion of Principal/Clinical Investigator or designated physicians, as judged by medical history) in the last 12 months
7. Have positive result of urine drug abuse testing on opioids (Mor, MTD), cannabinoids (THC), Meth, Coc or MDMA at screening visit or before dose administration at each period
8. Alcohol abuse or excessive use (in the opinion of Principal/Clinical Investigator or designated physicians, as judged by medical history) in the last 12 months
9. Have positive result of alcohol breathing test at screening visit or before dose administration at each period
10. Female subject is pregnant or breast feeding.
11. Difficulties fasting or consuming standard meals
12. Difficulties swallowing whole tablets
13. Donation or loss of whole blood:

    1. ≥50 mL and ≤499 mL within 30 days prior to Day 1
    2. ≥500 mL within 56 days prior to Day 1
14. Participation in any investigational drug study within 30 days from screening visit (from the last follow-up visit to the screening visit).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males and Females
Enrollment: 48 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Cmax | 4 months
  Peak Plasma Concentration
AUC | 4 months
  Area under the plasma concentration

SECONDARY OUTCOMES:
tmax | 4 months
  Time to reach Cmax
t1/2 | 4 months
  apparent terminal elimination half-life
λz | 4 months
  apparent terminal elimination rate constant
AUC0-t/AUC0-∞ | 4 months
  Ratio of Area under the curves
residual area | 4 months
  residual area

CONTACTS AND LOCATIONS:
Overall Officials: Ariya Khunvichai, Ph.D, Study Director — Medica Innova Co., Ltd.
Locations (1):
- Medica Innova Co Ltd, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No